CLINICAL TRIAL: NCT04145869
Title: Prospective Comparison of Intraoperative Fluorescent and X-ray Cholangiography for Visualisation of the Bile Duct Anatomy in Patients With Acute Cholecystitis
Brief Title: Fluorescent Cholangiography During Acute Cholecystitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Hillerod Hospital, Denmark (Other); Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Lars Lang Lehrskov, Principal investigator, Hvidovre University Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IFC3
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acute Cholecystitis
Keywords: Fluorescence; Cholangriography; Cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluorescent cholangiography (Experimental): Intraoperative fluorescent cholangiography using an intravenous injection of 5mg Indocyanine green
  Interventions: Procedure: Cholangiography
- X-ray cholangiography (Active Comparator): Intraoperative X-ray cholangiography using an intraductal (cystic duct) injection of Iohexol
  Interventions: Procedure: Cholangiography

INTERVENTIONS:
Procedure: Cholangiography — All patients will be subjected to intraoperative fluorescent and concommitant X-ray cholangiography

SUMMARY:
This study compares the visualizationrate of fluorescent and X-ray cholangiography during laparoscopic cholecystectomy for acute cholecystitis

ELIGIBILITY:
Inclusion criteria

* Patient scheduled for acute laparoscopic cholecystectomy due to acute cholecystitis with ≤ 5 days of complaints (in Denmark the national consensus for surgical window)

Exclusion criteria

* Laparoscopic operation converted to open operation prior to completed fluorescent and X-ray cholangiography
* Allergy towards iodine, Iohexol or indocyanine green
* Legally incompetent (any reason)
* Cholangitis (as defined above)15
* Withdrawal of inclusion consent at any time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visualizationrate | 1 hour
  Percentage of patients with visualization of the structure: the cystic duct - common hepatic duct - common bile duct junction.

SECONDARY OUTCOMES:
Visualizationrate | 1 hour
  Percentage of patients with visualization of the structure2: right and left hepatic ducts, common hepatic duct, common bile duct, cystic duct
Bile duct stones | 1 hour
  Percentage of patients with visualization of bile duct stones

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Northzealand Hospiral Hillerød, Hillerød, Danmark
  - Hvidovre University Hospital, Hvidovre, Danmark
  - Zealand University Hospital Køge, Køge

IPD SHARING:
Plan to Share IPD: Undecided